CLINICAL TRIAL: NCT03521817
Title: The Effects of Alcohol Consumption on Central Adiposity and Testosterone Following Weight Loss in Obese, Pre-menopausal Women
Brief Title: The Effects of Alcohol Consumption on Central Adiposity
Acronym: CONSUME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Ursula A. White (Unknown); Frank L. Greenway (Unknown); Martin, Corby, K., M.D. (Individual)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-057
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Alcohol Drinking; Weight Loss; Adiposity; Obesity; Visceral Obesity
MeSH Terms: conditions — Alcohol Drinking; Weight Loss; Obesity; Obesity, Abdominal | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This is a between-subjects parallel study design. All women will undergo a 30% energy restriction for 8-weeks and will be randomized to an ethanol-consuming group or a non-ethanol control group at the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol (Experimental): Etoh will have a 30% reduction in calories from weight maintenance and will consume the same percentage of each traditional macronutrient (20% protein, 50% carbohydrate, and 30% fat; (minus the ~240 kcals from ethanol). The Etoh group will consume a 30% energy restriction diet that will also include ~2.5 standard drinks, or 35 grams of ethanol, administered as 80-proof distilled spirits (e.g. 80 proof gin, rum, vodka, whiskey, or tequila).
  Interventions: Other: Alcohol
- No Alcohol (Active Comparator): No Etoh will have a 30% reduction in calories from weight maintenance and will consume the same percentage of each traditional macronutrient (20% protein, 50% carbohydrate, and 30% fat).
  Interventions: Other: No Alcohol

INTERVENTIONS:
Other: Alcohol — The ethanol group will consume a 30% energy restriction diet that will also include ~2.5 standard drinks, or 35 grams of ethanol, administered as 80-proof distilled spirits (e.g. 80 proof gin, rum, vodka, whiskey, or tequila). In the United States, one "standard" drink contains roughly 14 grams of pure alcohol.
  Other Names: Etoh
  Arms: Alcohol
Other: No Alcohol — This group will not consume alcohol. Thus 0 kcal/d will come from alcohol
  Other Names: No Etoh
  Arms: No Alcohol

SUMMARY:
The objective of the proposed study is to enroll women with obesity that will undergo a controlled, energy restricted feeding intervention to test the effects of chronic ethanol consumption on adipose distribution and circulating testosterone during weight loss.

DETAILED DESCRIPTION:
Alcohol (i.e. ethanol) is one of the most widely used recreational substances by humans and is consumed regularly by much of the U.S. population. Despite the high prevalence of alcohol intake, the metabolic health effects associated with use have not been firmly established. There is a paucity of data from longitudinal studies in humans that examine the metabolic response to routine alcohol consumption in a randomized controlled trial (RCT).

This is a novel pilot study to examine, for the first time, the effects of ethanol consumption on fat distribution and testosterone during weight loss in a RCT. Findings from this study would provide insight into an interesting and unanswered question -- does routine alcohol intake exert unfavorable health effects despite the expected beneficial outcomes of caloric restriction and weight loss? This research may provide new knowledge of the metabolic outcomes resulting from alcohol intake and pathways that may be involved leading to potential new therapeutic targets of treatment.

The objective of the proposed study is to enroll women with obesity that will undergo a controlled, energy restricted feeding intervention to test the effects of chronic ethanol consumption on adipose distribution and circulating testosterone during weight loss. Women will be randomized to an ethanol-free control group or an ethanol-consuming group, and all will consume 30% energy-restricted diets.

ELIGIBILITY:
Inclusion Criteria:

* - Pre-menopausal women only
* 21-40 years of age
* BMI 27-50 kg/m2 (+/- 0.5 will be accepted)
* Must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as double barrier methods [male condom with spermicide, with or without cervical cap or diaphragm], implants, intrauterine contraceptive devices, tubal ligation (surgically sterile), abstinence, or in an established relationship with a vasectomized or same sex partner) during the entire duration of the study
* Must be willing to adhere to all study procedures, including consumption of all study foods and beverages and attendance at all study visits
* - Must be willing to eat at least one meal at PBRC 3 times per week on weekdays (excluding holidays)
* Must be willing to consume alcohol
* Must be willing to abstain from alcohol for 8-weeks if randomized to non-alcohol control group.
* Must be a daily, or almost daily drinker, defined as typically consuming at least 8 drinks per week, but no more than 4 per day
* Must be willing to undergo an overnight alcohol test (at home) of ethanol at the proposed dose before enrollment in the study
* Must have access to a device that can be used for video monitoring of compliance (i.e. Skype)
* Must be willing to have your blood stored for future research

Exclusion Criteria:

* - Non-drinkers of alcohol
* Habitual binge drinkers, as defined by the consumption of ≥ 4 standard drinks per day or ≥ 28 drinks per week.
* Self-reported alcoholics or a history of alcoholism
* Have a 1st degree relative with alcoholism
* Any attendance or inpatient stay for alcohol or drug treatment
* Display any characteristics of current or future substance abuse disorders
* Presence of any psychiatric, behavioral, or medical disorder that, in the opinion of the PIs, Co-I, or MI, may interfere with study participation, the ability to adhere to the protocol, or has the potential for increased substance abuse
* Prescription medications that interact with alcohol intake
* Abnormal screening laboratory safety tests
* Smokers
* Diagnosis of Type 1 or 2 diabetes mellitus, cancer, or major organ disease
* Serious digestive disorders
* Conditions that affect metabolism or body weight (i.e. uncontrolled thyroid conditions, bariatric surgery, pregnancy, breastfeeding)
* Partial and/or full hysterectomy
* Hormonal pharmaceutical contraceptives including oral contraception (birth control pills), injectables (Depo-Provera), or the patch (Xulane)
* PCOS
* Use of medications that affect body weight or metabolism (i.e. atypical antipsychotics, weight loss medications).
* Not willing to store biospecimens for future use

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol | No Alcohol
Started | 7 | 5
Completed | 7 | 4 (1 completer was non adherent based on weekly intervention body weight)
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol | No Alcohol | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9) | 31 (7) | 32 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Central (Abdominal) Adiposity
Description: change in visceral abdominal adipose tissue from baseline to post intervention
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Alcohol | No Alcohol
Number analyzed (Participants) | 7 | 3
kg | -0.250 (0.115) | -0.071 (0.075)
Statistical Analysis 1: Comparison: Alcohol vs No Alcohol; Test type: Other; p < 0.231, t-test, 2 sided; Mean Difference (Net) = -0.18, Standard Error of Mean 0.14

ADVERSE EVENTS:
Time Frame: From baseline to completion of study 8 weeks later. Furthermore follow-up calls and emails (not in person visits) were performed post study. Thus total period of time adverse event data were collected was 12 weeks.
Arm/Group | Alcohol | No Alcohol
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 1/7 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcohol (N=7) | No Alcohol (N=5)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritis (itching) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory complaints (cold) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
One additional person was randomized due to a participant dropout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT03521817/Prot_000.pdf